CLINICAL TRIAL: NCT01315340
Title: Measurement of Ocular Rigidity, Outflow Facility and Ocular Blood Flow in Glaucomatous and Normal Eyes
Brief Title: Ocular Rigidity and Outflow Facility in Glaucomatous and Normal Eyes
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Larissa University Hospital (Other)
Collaborators: University of Crete (Other)
Responsible Party: Principal Investigator, Anna Dastiridou, MD, PhD, Larissa University Hospital
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 8068
Record Dates: First submitted 2011-03-09; First posted 2011-03-15 (Estimated); Last update posted 2022-08-16 (Actual); Status verified 2022-08

CONDITIONS: Glaucoma
MeSH Terms: conditions — Glaucoma | interventions — Intraocular Pressure

ARMS (2):
- Glaucoma Patients (Experimental)
  Interventions: Procedure: Ocular rigidity, outflow facility and intraocular pressure measurement
- Control subjects (Active Comparator)
  Interventions: Procedure: Ocular rigidity, outflow facility and intraocular pressure measurement

INTERVENTIONS:
Procedure: Ocular rigidity, outflow facility and intraocular pressure measurement — The measurement procedure includes cannulation of the anterior chamber of the eye, under sterile conditions. Infusion of the eye with microvolumes of a saline solution is performed, followed by manometric measurement of intraocular pressure, in order to quantify ocular rigidity. Outflow facility is estimated from recordings of intraocular pressure after the infusion is stopped.

SUMMARY:
Ocular rigidity characterizes the relationship between pressure and volume changes in the human eye and is expressed as a macroscopic coefficient. Outflow facility is a measure of the resistance of the conventional outflow pathway and represents a parameter that is of interest in glaucoma.

Difficulties in the measurement of ocular rigidity in the living human eye have limited our knowledge on this parameter. However, ocular biomechanics have been implicated in the pathogenesis of this disease. The aim of this study is to characterize the pressure volume relation and quantify ocular rigidity and outflow facility in glaucomatous and normal eyes. For this purpose, the investigators have recently developed a manometric method for the measurement of ocular rigidity and outflow facility.

ELIGIBILITY:
Inclusion Criteria:

* Patients with primary open or pseudoexfoliation glaucoma that are undergoing cataract surgery
* Patients undergoing cataract surgery without evidence of other ocular disease.

Exclusion Criteria:

* Evidence of any ocular disease, other than specified in the inclusion criteria
* Previous ophthalmic surgery or trauma
* Significant visual field defect (MD<-12dB) or an increased cup to disc ratio (>0.9).

Ages: 40 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2011-03; Primary Completion 2023-03 (Estimated); Study Completion 2024-07 (Estimated)

PRIMARY OUTCOMES:
Ocular rigidity coefficient | 2 minutes measurement of ocular rigidity
Outflow facility coefficient | 3-4 minutes measurement of outflow facility

SECONDARY OUTCOMES:
Ocular pulse amplitude | 6 minutes
Pulsatile ocular blood flow | 6 minutes

CONTACTS AND LOCATIONS:
Overall Officials: Ioannis Pallikaris, MD, Principal Investigator — University of Crete
Locations (1):
- Ophthalmology Department, University Hospital of Larissa, Larissa, Greece

REFERENCES:
- [Background] Dastiridou AI, Ginis HS, De Brouwere D, Tsilimbaris MK, Pallikaris IG. Ocular rigidity, ocular pulse amplitude, and pulsatile ocular blood flow: the effect of intraocular pressure. Invest Ophthalmol Vis Sci. 2009 Dec;50(12):5718-22. doi: 10.1167/iovs.09-3760. Epub 2009 Jul 15. PMID 19608534
- [Background] Pallikaris IG, Kymionis GD, Ginis HS, Kounis GA, Christodoulakis E, Tsilimbaris MK. Ocular rigidity in patients with age-related macular degeneration. Am J Ophthalmol. 2006 Apr;141(4):611-5. doi: 10.1016/j.ajo.2005.11.010. PMID 16564793
- [Background] Pallikaris IG, Kymionis GD, Ginis HS, Kounis GA, Tsilimbaris MK. Ocular rigidity in living human eyes. Invest Ophthalmol Vis Sci. 2005 Feb;46(2):409-14. doi: 10.1167/iovs.04-0162. PMID 15671262
- [Background] Dastiridou AI, Ginis H, Tsilimbaris M, Karyotakis N, Detorakis E, Siganos C, Cholevas P, Tsironi EE, Pallikaris IG. Ocular rigidity, ocular pulse amplitude, and pulsatile ocular blood flow: the effect of axial length. Invest Ophthalmol Vis Sci. 2013 Mar 1;54(3):2087-92. doi: 10.1167/iovs.12-11576. PMID 23462745
- [Background] Dastiridou AI, Tsironi EE, Tsilimbaris MK, Ginis H, Karyotakis N, Cholevas P, Androudi S, Pallikaris IG. Ocular rigidity, outflow facility, ocular pulse amplitude, and pulsatile ocular blood flow in open-angle glaucoma: a manometric study. Invest Ophthalmol Vis Sci. 2013 Jul 10;54(7):4571-7. doi: 10.1167/iovs.13-12303. PMID 23761082
- [Background] Karyotakis NG, Ginis HS, Dastiridou AI, Tsilimbaris MK, Pallikaris IG. Manometric measurement of the outflow facility in the living human eye and its dependence on intraocular pressure. Acta Ophthalmol. 2015 Aug;93(5):e343-e348. doi: 10.1111/aos.12652. Epub 2015 Feb 1. PMID 25645503